CLINICAL TRIAL: NCT03985059
Title: Impact of Verticalization on Intracranial Hemodynamics Assessed in Transcranial Doppler at the Acute Phase of Cerebral Infarction (STAND : iSchemic sTroke evAluated at Bed Side With ultrasouND)
Brief Title: Impact of Verticalization on Intracranial Hemodynamics Assessed in Transcranial Doppler at the Acute Phase of Cerebral Infarction
Acronym: STAND
Status: Terminated | Type: Observational
Why Stopped: no need to include more patients for analysis. 40 patients initially (36 actual)
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: MMI_2018_12
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Verticalization; Doppler; Intracranial hemodynamic; Cerebral artery velocity
MeSH Terms: conditions — Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients with ischemic stroke or transient ischemic attack who have carotid stenosis greater than 50% NASCET (North American Symptomatic Carotid Endarterectomy Trial) or an occlusion.
  Interventions: Other: Transcranial Doppler
- Controls: Patients with ischemic stroke or transient ischemic attack who do not have carotid stenosis greater than 50% NASCET (North American Symptomatic Carotid Endarterectomy Trial) or an occlusion.
  Interventions: Other: Transcranial Doppler

INTERVENTIONS:
Other: Transcranial Doppler — Initially, the patient will be placed in a strict supine position (at 0°) in his hospital bed in the USINV, according to the usual care. In a second step, the patient will be verticalized (from 0° to 90°). HI parameters in supine position and during verticalization will be recorded continuously by placing the transcranial Doppler helmet.
  After 15 minutes of recording, the patient will be placed back in supine position. The end of the patient's participation in the study will correspond to the removal of the helmet.

SUMMARY:
The management of patients with ischemic stroke or transient ischemic attack is based on the preservation of a brain area by maintaining sufficient intracranial hemodynamics (IH) and with rapid recanalization.

The impact of the patient's position (supine or seated position) on the IH in the event of narrowing or occlusion of an artery is poorly assessed but may be of particular importance. Variations in blood flow according to the positioning of the patient's body are measurable using a transcranial Doppler.

The main objective is to verify whether intracerebral hemodynamic changes during early verticalization after ischemic stroke or transient ischemic attack are more frequent in patients with carotid stenosis or occlusion compared to those without stenosis or occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke (AIC) or transient ischemic attack (AIT) of the carotid artery
* Duration of symptoms less than 48 hours
* Absence of homolateral or downstream intracranial stenosis or occlusion M1
* Lifting authorized by the referent clinician.
* Rankin's score before AIC/AIT ≤ 2

  • For cases:
* Carotid stenosis of more than 50% NASCET (North American Symptomatic Carotid Endarterectomy Trial) or an occlusion

  • For controls:
* Absence of carotid stenosis greater than 50% NASCET (North American Symptomatic Carotid Endarterectomy Trial) or occlusion

Exclusion Criteria:

- Disrupted vigilance

Secondary exclusion criteria:

* Absence of a homolateral temporal acoustic window at the lesion
* Impossibility to verticalize the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited during their hospitalization in the USINV for the management of ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a change in mean cerebral artery velocity (MCAVM) in transcranial Doppler | 2 minutes
  Percentage of patients with a change in mean cerebral artery velocity (MCAVM) in transcranial Doppler (defined by a variation of more than 10%) on the symptomatic side evaluated in transcranial Doppler when changing from the lying position (0°) to the 90° position (measured 2 minutes after verticalization).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmique Adolphe de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: No